CLINICAL TRIAL: NCT02315430
Title: A Phase II Trial of Cabozantinib (XL-184) (NSC #761968) in Women With Recurrent, Clear Cell Carcinoma of the Ovary, Fallopian Tube, or Peritoneum
Brief Title: Cabozantinib-S-Malate in Treating Patients With Recurrent or Progressive Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02411; NCI-2014-02411 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY001 (Other: NRG Oncology); NRG-GY001 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Ovarian Clear Cell Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cabozantinib-s-malate) (Experimental): Patients receive cabozantinib-s-malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL184
Other: Laboratory Biomarker Analysis — Optional correlative studies

SUMMARY:
This phase II trial studies how well cabozantinib-s-malate works in treating patients with ovarian, fallopian tube, or primary peritoneal cavity cancer that has come back or is growing, spreading, or getting worse. Cabozantinib-s-malate may stop the growth of tumor cells by blocking the growth of new blood vessels necessary for tumor growth and also by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the anti-tumor activity of cabozantinib (XL184) (cabozantinib-s-malate) in women with persistent or recurrent clear cell ovarian cancer, based on the proportion of patients who survive progression-free for at least 6 months and the proportion who have objective tumor response (complete or partial).

SECONDARY OBJECTIVES:

I. To determine the nature, frequency and maximum degree of toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v)4 for cabozantinib (XL184).

II. To determine the progression free survival (PFS) and overall survival (OS) for patients with persistent or recurrent clear cell ovarian cancer treated with cabozantinib (XL184).

TERTIARY OBJECTIVES:

I. To examine the expression of phosphatase and tensin homolog gene (PTEN), phosphorylated v-akt murine thymoma viral oncogene homolog 1 (pAKT), cyclin E, and met proto-oncogene (MET) in formalin-fixed, paraffin-embedded tumor.

II. To examine MET amplification (fluorescence in situ hybridization) in tumor specimens and the relationship to response.

OUTLINE:

Patients receive cabozantinib-s-malate orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* A retrospective review of all patients entered will be performed to confirm clear cell histology; patients must have recurrent or, progressive clear cell ovarian cancer not solely based on cancer antigen (CA)-125; primary tumors must be at least 50% clear cell histomorphology in order to be eligible or have a histologically documented recurrence with at least 50% clear cell histomorphology; recurrence should be biopsy proven unless the tumor is located in an area deemed unsafe to biopsy by the surgeon; if a biopsy can be obtained without significant risk, then biopsy should be obtained
* If the primary tumor had at least 50% clear cell histomorphology, a biopsy of the recurrent or persistent tumor is not required; the percentage of clear cell histomorphology must be documented in the pathology report or in an addendum to the original report; if slides of the primary tumor are not available for review due to disposal of slides by the histology laboratory (typically 10 years after diagnosis), biopsy of recurrent or persistent disease is required
* If slides of the primary tumor are not available for review, a biopsy of the recurrent or persistent tumor is required to confirm at least 50% clear cell histomorphology; the percentage of involvement must be documented in the pathology report or in an addendum to the original report
* All patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* All patients must submit unstained slides of primary or recurrent tumor for translational analysis
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease; platinum sensitive and resistant patients are eligible
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease
* Concomitant use of additional anti-neoplastic agents will not be allowed in this study
* Patients may not have received previous therapy with a MET inhibitor
* Patients must not be eligible for a higher priority (e.g.; phase II/III), National Surgical Adjuvant Breast and Bowel Project, Radiation Therapy Oncology Group, and Gynecologic Oncology Group (NRG) protocol for the same population if one exists
* Patients must be recovered from effects of recent surgery (28 days must elapse between surgery and the start of treatment with cabozantinib)
* Patients must have >= 4 weeks since prior chemotherapy or radiation (>= 6 weeks for nitrosoureas or mitomycin C)
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination within 28 days prior to registration
* The trial is open only to women with recurrent, progressive clear cell carcinoma of the ovary
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (Karnofsky >= 60%) within 28 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Leukocytes >= 3,000/mcL
* Hemoglobin >= 9 g/dL
* Serum albumin >= 2.8 g/dL
* Prothrombin time (PT) such that international normalized ratio (INR) is less than or equal to 1.3 x upper limit of normal (ULN)
* Partial thromboplastin time (PTT) less than or equal to 1.3 x ULN
* Creatinine less than or equal to 1.5 times the ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The urine protein: creatinine ratio (UPCR) is derived as follows: protein concentration (mg/dL)/creatinine (mg/dL); patients must have a UPCR < 1.0 to allow participation in the study
* Bilirubin less than or equal to 1.5 ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 times the ULN, unless subjects have liver metastasis, in which case both AST and ALT must be less than or equal to 5 times the ULN
* Lipase less than or equal to 2 x ULN
* No clinical evidence of pancreatitis
* Patients must have a normal baseline thyroid stimulating hormone (TSH); a history of hypothyroidism and/or hyperthyroidism is allowed
* Women of childbearing potential must have a negative pregnancy test at screening; women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal; post-menopause is defined as amenorrhea >= 12 consecutive months; note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, ovarian suppression or any other reversible reason; women should stop breastfeeding while participating in this trial; male partners of women participants should also use medically-acceptable forms of contraception during the study
* The patient must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Human immunodeficiency virus (HIV) positive patients
* Patients with serious non-healing wound, ulcer, or bone fracture
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel); low dose aspirin (=< 81 mg/day), low-dose warfarin (=< 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within 6 months of the first date of treatment on this study
* Patients with clinically significant cardiovascular disease; this includes:

  * Poorly controlled hypertension (> 140 mm Hg and > 90 mm Hg for systolic and diastolic blood pressure [BP]) are ineligible
  * Myocardial infarction or unstable angina within 6 months prior to registration; New York Heart Association (NYHA) grade II or greater congestive heart failure
  * Cardiac arrhythmia requiring medication
* Grade II or greater peripheral vascular disease based on National Cancer Institute (NCI) Common Toxicity Criteria (CTC); e.g. ischemic rest pain, minor tissue loss, and ulceration or gangrene
* Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medication are ineligible; patients with a history of hypothyroidism are eligible provided they are currently euthyroid
* Patients who have a major surgical procedure, or significant traumatic injury within 28 days prior to the first date of treatment on this study, or anticipation of need for major surgical procedure during the course of the study; patients with placement of vascular access device or core biopsy within 7 days prior to the first date of treatment on this study
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy
* Patients must not be eligible for a higher priority NRG clear cell protocol (Gynecologic Oncology Group [GOG]-0283); rare patients ineligible for GOG-0283 may be eligible for this trial without prior treatment on dasatinib therapy (e.g. they have been deemed allergic to dasatinib)
* Patients who cannot swallow pills

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-02-09 (Actual); Study Completion 2019-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Farley, Principal Investigator — NRG Oncology
Locations (410):
- United States (410):
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arizona Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Monongalia Hospital, Morgantown, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 4/1/2015 and closed to accrual on 10/31/2016.
Groups:
- Cabozantinib: Cabozantinib (XL184) 60 mg once a day continuously, repeated in 4 week cycles until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | Cabozantinib
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Who Survive Progression Free for at Least 6 Months
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression was based on RECIST 1.1. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Every 8 weeks during treatment, assessesd up to 6 months for progression free survival.
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 13
percentage of participants | 23 [7 to 49]

2. Primary Outcome: Objective Tumor Response
Description: Complete and Partial Tumor Response by RECIST 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Every 8 weeks during treatment;assessed up to 20 months.
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 13
percentage of participants | 0 [0 to 21]

3. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: Grade 3 or higher adverse events were graded by CTC AE v 4.
Time Frame: Every cycle while on treatment, up to 30 days after treatment ends, an average of 14 months.
Population: Eligible and Treated Patients
Measure: Number; unit: participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 13
participants
  Nausea | 3
  Vomiting | 3
  Thromboembolic Event | 3
  Fatigue | 2
  Dehydration | 2
  Dyspnea | 2
  Abdominal Pain | 1
  Diarrhea | 1
  Gastrointestinal Pain | 1
  Pain | 1
  Alanine aminotransferase increased | 1
  Alkaline phosphatase increased | 1
  Platelet count decreased | 1
  Hypoalbuminemia | 1
  Hyponatremia | 1
  Back pain | 1
  Bone pain | 1
  Syncope | 1
  Pleural effusion | 1
  Hypertension | 1

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression was based on RECIST 1.1
Time Frame: Tumor scan done every 8 weeks during treatment, Average progression free survival was 3.6 months.
Population: Eligible and Treated Patients
Measure: Mean (90% Confidence Interval); unit: months
Arm/Group | Cabozantinib
Number analyzed (Participants) | 13
months | 3.6 [1.8 to 7.9]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, up to 20.1 months.
Population: Eligible and Treated Patients
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cabozantinib
Number analyzed (Participants) | 13
Months | 8.1 [2.7 to NA] — Length of overall survival was not reached at time of analysis, but is >20.1 months

ADVERSE EVENTS:
Time Frame: Study Treatment and up to 30 days after study treatment an average of 14 months.
Arm/Group | Cabozantinib
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=13)
Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic Event (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=13)
Anemia (Blood and lymphatic system disorders) | 5
Ventricular Tachycardia (Cardiac disorders) | 1
Chest Pain - Cardiac (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Floaters (Eye disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 8
Bloating (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 7
Mucositis Oral (Gastrointestinal disorders) | 7
Oral Pain (Gastrointestinal disorders) | 3
Abdominal Distension (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 10
Pancreatitis (Gastrointestinal disorders) | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Pain (General disorders) | 3
Fatigue (General disorders) | 11
Fever (General disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Weight Loss (Investigations) | 5
Weight Gain (Investigations) | 1
Platelet Count Decreased (Investigations) | 2
Lipase Increased (Investigations) | 4
Creatinine Increased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 1
Cardiac Troponin I Increased (Investigations) | 1
Blood Bilirubin Increased (Investigations) | 1
White Blood Cell Decreased (Investigations) | 2
Aspartate Aminotransferase Increased (Investigations) | 7
Alkaline Phosphatase Increased (Investigations) | 7
Alanine Aminotransferase Increased (Investigations) | 5
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 6
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2
Memory Impairment (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 8
Syncope (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Skin Induration (Skin and subcutaneous tissue disorders) | 1
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 3
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Thromboembolic Event (Vascular disorders) | 5
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 6
Flushing (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT02315430/Prot_SAP_000.pdf